CLINICAL TRIAL: NCT02608658
Title: Evaluation of Serum-Derived Bovine Immunoglobulin Protein Isolate in Subjects With Decompensated Cirrhosis With Ascites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: American College of Gastroenterology (Other); Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Muhammad Hammami, MD, Housestaff Resident, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: StLouisU 25320
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Cirrhosis of the Liver; Ascites; Spontaneous Bacterial Peritonitis
Keywords: Cirrhosis; Ascites; SBP
MeSH Terms: conditions — Fibrosis; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional Arm (Experimental): The experimental arm of this study will involve all patients in this study. Subjects will be evaluated in a clinical setting and undergo a brief healthcare questionnaire, blood work, and a breath test. Subjects will then take a medical food (EnteraGam) twice daily for 8 weeks total, after which they will be seen in clinic at 4 weeks for follow up and then at 8 weeks to repeat the healthcare questionnaire, breath tests, and blood draw.
  Interventions: Other: Medical food, EnteraGam (Serum-Derived Bovine Immunoglobulin)

INTERVENTIONS:
Other: Medical food, EnteraGam (Serum-Derived Bovine Immunoglobulin) — Visit 1, screening (Day 0): At this visit, the investigators of the study will:
  * Obtain demographic information, as will past medical history and medications.
  * Perform a physical examination.
  * Collect samples for labs
  * Administer the Chronic Liver Disease Questionnaire (CLDQ)
  * Perform a lactulose breath test
  From Day 0 to 8 weeks: subjects will take the medical food twice daily
  Visit 2, Week 4 (Day 28 +/- 3): At this visit, the investigators of the study will:
  * Perform a physical examination
  * Collect and record returned investigational product
  * Dispense investigational product and instruct again regarding use
  * Record any adverse events
  Visit 3, Week 8 (Day 56 +/- 3): At this visit, the investigators of the study will:
  * Perform a physical examination.
  * Collect samples for labs
  * Administer the Chronic Liver Disease Questionnaire (CLDQ)
  * Perform a lactulose breath test
  Other Names: Serum-Derived Bovine Immunoglobulin

SUMMARY:
This protocol represents an open-label pilot study to assess whether oral administration of SBI in subjects with decompensated cirrhosis with ascites can lead improvements in the management of the disease. The impact of SBI therapy will be based on changes to markers of bacterial translocation, gut barrier damage, and inflammation as well as the impact on rates of SIBO. Study subjects will be given one packet of EnteraGam, each packet containing 5.0 g SBI, twice daily for 8 weeks.

DETAILED DESCRIPTION:
The Gut Barrier and Pathological Bacterial Translocation: The "Achilles Heel" of Hepatology

The intestinal wall is a complex barrier that exists between humans and their environment. Inside the intestinal lumen, the commensal flora exposes the epithelium to nearly 100 trillion bacteria.1 This epithelial layer provides a surface area of 400 square meters, lined with tight junctions that prevent the translocation and paracellular transport of luminal antigens including bacteria.2 In addition to this mechanical barrier, the wall of the intestine is lined with mucosal immune defenses, notably gut-associated lymphoid tissue (GALT), the largest immunologic organ in the body.1 Under normal circumstances, this functional and efficient barrier prevents entry of bacteria from the outside world.

Failure of this intestinal barrier, along with an increased rate of pathological bacterial translocation, has been shown to be associated with increasing severity of liver disease and the development of decompensated cirrhosis.3 Factors thought to contribute to bacterial translocation in subjects with cirrhosis include small intestinal bacterial overgrowth (SIBO), which is known to have an increased prevalence in subjects with cirrhosis compared to those without4, hyperdynamic portal status, alterations in the GALT tissue altering the immune response, and impaired intestinal permeability seen in subjects with ascites.3 This increased permeability is believed to result from structural abnormalities in the intestinal mucosa, including widening of intercellular spaces, edema, inflammation, and vascular congestion.5-7

Failure of the intestinal barrier is routinely thought to play an important role in the natural course of cirrhosis, so much so that this has been referred to as hepatology's "Achilles heel."8 Pathologic bacterial translocation across the intestinal epithelium is suspected to impact the clinical course of liver cirrhosis by triggering encephalopathy, hepatic failure, and hepatorenal syndrome, in addition to having a long known role as an underlying mechanism of the development of spontaneous bacterial peritonitis (SBP) and other bacterial infections in this population.9 Given that SBP is associated with high mortality rates ranging from 10-42%,10 and that subjects with cirrhosis have increased susceptibility to infections, antibiotic prophylaxis has emerged as a widely accepted strategy in subjects at increased risk for bacterial translocation, such as those with active gastrointestinal bleeding and low protein content ascites. However, this therapeutic strategy has the potential of selecting resistant bacterial strains and increasing the risk of subjects developing Clostridium difficile associated diarrhea.

Alternative methods for the prevention of SBP and bacterial infections in subjects with cirrhosis could prove to be very beneficial in reducing mortality and preventing the development of antibiotic resistance. In particular, preventing pathological bacterial translocation at the intestinal barrier could be highly effective.

Serum-Derived Bovine Immunoglobulin: a Logical Therapy to Improve Gut Barrier Function

Immunoglobulins taken orally are known to play a prominent role in health and development given the known benefits of human milk and colostrum, a form of milk produced by mammals which contains significant amounts of antibodies.11 Recognition of the essential nature of these antibodies led to the development of commercial plasma-derived protein concentrates containing immunoglobulins, which have been used for decades in animal husbandry to promote growth and manage intestinal inflammation in immune-compromised young animals.12-14

Serum-derived bovine immunoglobulin / protein isolate (SBI) is a novel medical food marketed under the brand name, EnteraGam®. This product is currently indicated (see EnteraGam package insert for details) for the clinical dietary management of several forms of enteropathy, including diarrhea predominant irritable bowel syndrome (IBS-D) and intestinal bowel disease (IBD). While the term, enteropathy, refers to any pathology or disease of the intestines, known histological features can include blunting of intestinal villi, increased intra-epithelial lymphocytes causing reduced absorptive capacity, and increased gut permeability.12 In cases of enteropathy, a combination of factors including altered gut microbiota, increased intestinal inflammation, and worsening gut barrier dysfunction are known to increase the risk of bacterial translocation.12 Each of these factors is a potential target for SBI. In terms of altered gut microbiota, extensive literature has demonstrated broad bacterial antigen neutralizing capacity of ingested immunoglobulins.15-17 Likewise, many non-clinical studies have shown that SBI can reduce intestinal inflammation by decreasing mucosal cytokines and dampening immune activation.18-19 Furthermore, the available data suggest that oral immunoglobulin therapy benefits tight-junction integrity in epithelial barriers, as evidenced through increased transepithelial electrical resistance and reduction in radiolabeled 14C-inulin permeability across the intestine.19

To date, there is a large body of evidence showing that serum- or plasma-derived bovine immunoglobulin preparations can effectively manage the symptoms and harmful effects of enteropathy in both animals and humans. Animal studies include data regarding barrier function and nutrient absorption in animals including mice, rats, and pigs.12 Studies performed in children show promising results in terms of weight gain and the underlying problem of malabsorption.22-23 Among adults, preliminary studies show promising results of SBI in the management of HIV enteropathy in addition to diarrhea-predominant Irritable Bowel Syndrome.24,25 Collectively, there is strong evidence to support the theory that ingestion of oral immunoglobulins such as SBI could reduce the risk of bacterial translocation in patients with cirrhosis, namely by neutralizing bacterial antigen in the intestine, reducing intestinal inflammation, and decreasing permeability of the gut barrier.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have signed and dated an Institutional Review Board (IRB) approved informed consent form (ICF) prior to beginning any study-related activities
* Subjects will be males and females between the ages of 18 to 70 years (inclusive)
* Subjects must have a confirmed diagnosis of cirrhosis as determined by radiographical (presence of a nodular appearing liver on imaging), clinical (must have documentation from a provider and information verified independently by chart review), or histological evidence (presence of bridging fibrosis on a prior biopsy)
* Subjects must have ascites based off of clinical or radiographical evidence
* Subjects with a Model for End-Stage Liver Disease (MELD) score of less than 17 as documented by most recent lab results. Subjects must be capable of understanding the requirements of the study, be willing to comply with all the study procedures, and be willing to attend all study visits.
* Females of childbearing (reproductive) potential must have a negative pregnancy test at screening and agree to use an acceptable method of contraception throughout their participation in the study. Acceptable methods of contraception include:

  * double barrier methods (condom with spermicidal jelly or a diaphragm with spermicide),
  * hormonal methods (e. g. oral contraceptives, patches or medroxyprogesterone acetate), or
  * an intrauterine device (IUD) with a documented failure rate of less than 1% per year.
  * Abstinence or partner(s) with a vasectomy may be considered an acceptable method of contraception at the discretion of the investigator.

NOTE: Female subjects who have been surgically sterilized (e.g. hysterectomy or bilateral tubal ligation) or who are postmenopausal (total cessation of menses for >1 year) will not be considered "females of childbearing potential".

Exclusion Criteria:

* Subjects with a MELD score of 17 or greater as documented by most recent lab results, within 45 days of their consent date.
* Subjects with a history of TIPS (transjugular intrahepatic portosystemic shunt) placement
* Subjects with a history of inflammatory bowel disease
* Subjects who have signs and symptoms of active infection, such as fever (temperature greater than 100.4oF) or meeting criteria for Systemic Inflammatory Response Syndrome (defined as two of the following four:

  * (1) a temperature greater than 100.4oF,
  * (2) heart rate of greater than 90 beats per minute,
  * (3) respiratory rate greater than 20 breaths per minute, or
  * (4) leukocytosis or leukopenia defined as a WBC greater than 12,000 cells/mm3 or less than 4,000 cells/mm3).
* Subjects who are on chronic antibiotics for any reason (including for prophylaxis of SBP or hepatic encephalopathy)
* Subjects who have a history of hepatic encephalopathy requiring daily lactulose or daily rifaximin for therapy
* Subjects who have active substance abuse or psychiatric disorders felt to preclude the ability to complete this study, including any drug abuse and active alcohol use greater than 1 drink daily
* Subjects who have a poorly controlled medical condition that is felt to interfere with study procedures
* Subjects who have a known allergy or hypersensitivity to beef or any component of SBI
* Subjects who are pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change in Markers of Bacterial Translocation | At the start and end of the study (time 0 and at time 8 weeks) for each individual patient, the following labs will be drawn and assessed for change
  * LBP (Lipopolysaccharide binding protein)
  * Soluble CD14
  * Procalcitonin
  * high sensitivity C-Reactive Protein (CRP)
  * Intestinal Fatty Acid Binding Protein (I-FABP)

SECONDARY OUTCOMES:
Change in the prevalence of Small Intestinal Bacterial Overgrowth | At the start and end of the study (time 0 and at time 8 weeks) for each individual patient
  Hydrogen breath test (using lactulose as the substrate)
Change to Quality of Life | At the start and end of the study (time 0 and at time 8 weeks) for each individual patient
  Quality of life will be determined with the use of the Chronic Liver Disease Questionnaire (CLDQ), a validated questionnaire used in subjects with cirrhosis. The CLDQ includes 29 questions in six domains: abdominal symptoms (three questions), fatigue (five questions), systemic symptoms (five questions), activity (three questions), emotional function (eight questions), and worry (five questions).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hummami, MD, Principal Investigator — Saint Louis University Division of Gastroenterology
Locations (1):
- Saint Louis University Salus Center, GI/Hepatology Clinical Studies Unit, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No